CLINICAL TRIAL: NCT00364351
Title: A Phase III, International, Randomised, Double Blind, Parallel-Group Study to Assess the Efficacy of Zactima™ Versus Tarceva® in Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer After Failure of at Least One Prior Chemotherapy
Brief Title: Efficacy Trial Comparing ZD6474 With Erlotinib in NSCLC After Failure of at Least One Prior Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D4200C00057; EUDRACT No. 2006-000259-16
Record Dates: First submitted 2006-08-14; First posted 2006-08-15 (Estimated); Results first posted 2011-05-24 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non Small Cell Lung Cancer; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — vandetanib; Erlotinib Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Active Comparator): Erlotinib
  Interventions: Drug: Erlotinib
- 2 (Experimental): Vandetanib
  Interventions: Drug: Vandetanib

INTERVENTIONS:
Drug: Vandetanib — once daily oral tablet
  Other Names: ZD6474; ZACTIMA™
  Arms: 2
Drug: Erlotinib — oral dose
  Other Names: Tarceva®
  Arms: 1

SUMMARY:
To determine if ZD6474 a new investigational drug, is effective in treating Non Small Lung Cancer and if so, how it compares with another type of anti cancer therapy chemotherapy, Erlotinib

ELIGIBILITY:
Inclusion Criteria:

* Confirmed locally advanced or metastatic NSCLC
* Failure of at least one but not more than two prior chemotherapy regimens

Exclusion Criteria:

* Prior treatment with erlotinib (Tarceva), gefitinib (IRESSA), sunitinib (Sutent), sorafenib (Nexavar)
* Chemotherapy or other type of anti cancer therapy within 4 weeks of study start

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1574 (Actual)
Dates: Start 2006-08; Primary Completion 2008-09 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (153):
- United States (29):
  - Research Site, Berkeley, California
  - Research Site, Los Angeles, California
  - Research Site, Santa Rosa, California
  - Research Site, Boynton Beach, Florida
  - Research Site, Fort Myers, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Port Saint Lucie, Florida
  - Research Site, Wichita, Kansas
  - Research Site, Lexington, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Metairie, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Columbia, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Latham, New York
  - Research Site, Hickory, North Carolina
  - Research Site, Canton, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Greenville, South Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Amarillo, Texas
  - Research Site, Garland, Texas
  - Research Site, Webster, Texas
  - Research Site, Fairfax, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Burien, Washington
  - Research Site, Yakima, Washington
- Argentina (6):
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Córdoba
  - Research Site, Manuel B. Gonnet
  - Research Site, Ramos Mejía
  - Research Site, Rosario
  - Research Site, Santa Fe
- Australia (9):
  - Research Site, Ashford
  - Research Site, Bedford Park
  - Research Site, Chermside
  - Research Site, Geelong
  - Research Site, Hornsby
  - Research Site, Kogarah
  - Research Site, Malvern
  - Research Site, Prahran
  - Research Site, Wodonga
- Brazil (7):
  - Research Site, Belo Horizonte
  - Research Site, Caxias do Sul
  - Research Site, Curitiba
  - Research Site, Goiânia
  - Research Site, Porto Alegre
  - Research Site, Santo André
  - Research Site, São Paulo
- Canada (12):
  - Research Site, Kelowna, British Columbia
  - Research Site, Vancouver, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Oshawa, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Sault Ste. Marie, Ontario
  - Research Site, Thunder Bay, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, York, Ontario
  - Research Site, Charlottetown, Prince Edward Island
  - Research Site, Laval, Quebec
  - Research Site, Montreal, Quebec
- China (8):
  - Research Site, Beijing
  - Research Site, Dalian
  - Research Site, Hangzhou
  - Research Site, Nanjing
  - Research Site, Nanning
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Wuhan
- Denmark (3):
  - Research Site, Herlev
  - Research Site, København Ø
  - Research Site, Næstved
- France (6):
  - Research Site, Caen
  - Research Site, Clermont-Ferrand
  - Research Site, Marseille
  - Research Site, Paris
  - Research Site, Rennes
  - Research Site, Vesoul
- Germany (9):
  - Research Site, Göttingen
  - Research Site, Großhansdorf
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, Karlsruhe
  - Research Site, Löwenstein
  - Research Site, Mainz
  - Research Site, Mönchengladbach
  - Research Site, Ulm
- Research Site, Hong Kong, Hong Kong
- India (5):
  - Research Site, Bangalore
  - Research Site, Karnataka
  - Research Site, New Delhi
  - Research Site, Pune
  - Research Site, Trivandrum
- Indonesia (3):
  - Research Site, Bandung
  - Research Site, Jakarta
  - Research Site, Solo
- Italy (11):
  - Research Site, Ancona
  - Research Site, Avellino
  - Research Site, Catania
  - Research Site, Genova
  - Research Site, Mantova
  - Research Site, Milan
  - Research Site, Orbassano
  - Research Site, Parma
  - Research Site, Perugia
  - Research Site, Roma
  - Research Site, Rozzano
- Mexico (6):
  - Research Site, Juchitán
  - Research Site, Monterrey
  - Research Site, Morelia
  - Research Site, Puebla City
  - Research Site, Saltillo
  - Research Site, Zacatecas City
- Netherlands (4):
  - Research Site, Harderwijk
  - Research Site, Nieuwegein
  - Research Site, Rotterdam
  - Research Site, Zwolle
- Norway (7):
  - Research Site, Bergen
  - Research Site, Haugesund
  - Research Site, Kristiansand
  - Research Site, Oslo
  - Research Site, Stavanger
  - Research Site, Tromsø
  - Research Site, Trondheim
- Philippines (5):
  - Research Site, Cebu City
  - Research Site, Davao City
  - Research Site, Manila
  - Research Site, Pasay
  - Research Site, Quezon City
- Research Site, Seoul, South Korea
- Spain (6):
  - Research Site, Elche(Alicante)
  - Research Site, Jaén
  - Research Site, Madrid
  - Research Site, Mataró(Barcelona)
  - Research Site, Málaga
  - Research Site, Pamplona
- Taiwan (4):
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (4):
  - Research Site, Bangkok
  - Research Site, Chiang Mai
  - Research Site, Lampang
  - Research Site, Songkhla
- United Kingdom (7):
  - Research Site, Birmingham
  - Research Site, Cambridge
  - Research Site, Leicester
  - Research Site, Liverpool
  - Research Site, Nottingham
  - Research Site, Sheffield
  - Research Site, Wolverhampton

REFERENCES:
- [Result] Natale RB, Thongprasert S, Greco FA, Thomas M, Tsai CM, Sunpaweravong P, Ferry D, Mulatero C, Whorf R, Thompson J, Barlesi F, Langmuir P, Gogov S, Rowbottom JA, Goss GD. Phase III trial of vandetanib compared with erlotinib in patients with previously treated advanced non-small-cell lung cancer. J Clin Oncol. 2011 Mar 10;29(8):1059-66. doi: 10.1200/JCO.2010.28.5981. Epub 2011 Jan 31. PMID 21282542
- [Derived] Mishina A, Zhudenkov K, Helmlinger G, Peskov K. A Systematic Comparative Analysis of Tumor Size Models Based on Erlotinib Clinical Data in Advanced NSCLC. CPT Pharmacometrics Syst Pharmacol. 2025 Dec;14(12):1970-1981. doi: 10.1002/psp4.70095. Epub 2025 Aug 11. PMID 40785488
- [Derived] Platt A, Morten J, Ji Q, Elvin P, Womack C, Su X, Donald E, Gray N, Read J, Bigley G, Blockley L, Cresswell C, Dale A, Davies A, Zhang T, Fan S, Fu H, Gladwin A, Harrod G, Stevens J, Williams V, Ye Q, Zheng L, de Boer R, Herbst RS, Lee JS, Vasselli J. A retrospective analysis of RET translocation, gene copy number gain and expression in NSCLC patients treated with vandetanib in four randomized Phase III studies. BMC Cancer. 2015 Mar 23;15:171. doi: 10.1186/s12885-015-1146-8. PMID 25881079
- See also: Vandetanib_study_57_ZEST_CSP_redacted_SECURE — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=347&filename=Vandetanib_study_57_ZEST_CSP_redacted_SECURE.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled 24 August 2006, last patient enrolled 31 October 2007, cut off date 26 September 2008. 1574 patients were enrolled in the study.
Pre-assignment Details: 1574 patients were enrolled/screened to the study but only 1240 patients were entered treatment/randomized.
Groups:
- Vandetanib: Vandetanib 300 mg tablet taken once daily plus a placebo for erlotinib
- Erlotinib: Erlotinib 150 mg tablet taken once daily plus a placebo for vandetanib
Period: Overall Study
Arm/Group | Vandetanib | Erlotinib
Started | 623 (randomised patients) | 617 (randomised patients)
Completed | 31 (Ongoing study treatment at data cut-off date 26 Sep 2008.) | 34 (Ongoing study treatment at data cut-off date 26 Sep 2008.)
Not Completed | 592 | 583
Not completed — Adverse Event | 90 | 44
Not completed — Condition under investigation worsened | 469 | 497
Not completed — Prohibited concomitant medication | 0 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 30 | 29
Not completed — Incorrect enrollment | 1 | 1
Not completed — Sponsor decision | 1 | 0
Not completed — Poor treatment compliance | 0 | 3
Not completed — Investigator error | 0 | 2
Not completed — Patient could not travel to site | 0 | 1
Not completed — Randomised treatment not started | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Vandetanib: Vandetanib 300 mg
- Erlotinib: Erlotinib
- Total: Total of all reporting groups
Arm/Group | Vandetanib | Erlotinib | Total
Number analyzed (Participants) | 623 | 617 | 1240
Age, Continuous [Mean (Full Range); unit: years] | 60 [26 to 92] | 61 [26 to 85] | 60 [26 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 242 | 224 | 466
  Male | 381 | 393 | 774

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: Median time (in weeks) from randomisation until objective disease progression or death (by any cause in the absence of objective progression) provided death is within 3 months from the last evaluable Response Evaluation Criteria In Solid Tumors (RECIST) assessment.
  Progression was derived according to RECIST 1.0 and is defined as an increase of at least 20% in the total tumour size of measurable lesions over the nadir measurement, unequivocal progression in the non-target lesions or the appearance of one or more new lesions.
Time Frame: progressionRECIST tumour assessments carried out every 4 weeks up to week 16 then every 8 weeks thereafter from randomisation until the date of first documented objective disease progression or date of death from any cause, whichever came first, assessed.
Measure: Median (Full Range); unit: Weeks
Arm/Group | Vandetanib | Erlotinib
Number analyzed (Participants) | 623 | 617
Weeks | 11.3 [0.14 to 75.43] | 8.9 [0.43 to 80.43]

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from date of randomization until death. Any patient not known to have died at the time of analysis will be censored based on the last recorded date on which the patient was known to be alive (ie their status must be known at the censored date and should not be lost to follow up or unknown).
Time Frame: Time to death in months
Measure: Median (Full Range); unit: Months
Arm/Group | Vandetanib | Erlotinib
Number analyzed (Participants) | 623 | 617
Months | 6.9 [0.03 to 18.46] | 7.8 [0.10 to 20.04]

3. Secondary Outcome: Objective Response Rate (ORR)
Description: The ORR is the number of patients that are responders ie those patients with a confirmed best objective response of complete response (CR) or partial response (PR) as determined according to RECIST 1.0. CR is defined as the disappearance of all target lesions with no evidence of tumour elsewhere and PR is defined as at least a 30% reduction in the total tumour size of measurable lesions with no new lesions and no progression in the non-target lesions.
Time Frame: RECIST tumour assessments every 4 weeks up to week 16 then every 8 weeks thereafter from randomisation until the date of first documented objective disease progression or date of death from any cause, whichever came first, assessed up to 21 months
Measure: Number; unit: Participants
Arm/Group | Vandetanib | Erlotinib
Number analyzed (Participants) | 623 | 617
Participants | 75 | 74

4. Secondary Outcome: Disease Control Rate (DCR)
Description: Disease control rate is defined as the number of patients who achieved disease control at least 8 weeks following randomisation. Disease control is defined as a best objective response of complete response (CR), partial response (PR) or stable disease (SD) >= 8 weeks as determined according to RECIST 1.0. CR is defined as the disappearance of all target lesions with no evidence of tumour elsewhere, PR is defined as at least a 30% reduction in the total tumour size of measurable lesions with no new lesions and no progression in the non-target lesions and SD >= 8 is assigned to patients who have not responded and have no evidence of progression at least 8 weeks after randomisation.
Time Frame: RECIST tumour assessments carried out every 4 weeks until week 16 then every 8 weeks thereafter (+/- 3 days) from randomisation until objective progression
Measure: Number; unit: Participants
Arm/Group | Vandetanib | Erlotinib
Number analyzed (Participants) | 623 | 617
Participants | 254 | 242

5. Secondary Outcome: Time to Deterioration of Disease-related Symptoms (TDS) by EORTC Quality of Life Questionnaire - Pain
Description: Pain was assessed as the average score of two items: Question 9 ("Have you had pain") and 19 ("Did pain interfere with your daily activities") of the QLQ-C30.
  Time to deterioration in symptoms is defined as the interval from the date of randomization to the first assessment of worsened without an improvement in the next 28 days. A patient is defined as having a deterioration in symptoms if they have a single visit assessment of 'worsened' with no visit assessment of 'improved' within the next 28 days.
Time Frame: Disease-related symptom assessments are to be administered at screening (within 7 days before the first dose of study medication), every 4 weeks thereafter, at discontinuation of study treatment and at the 30-day follow-up visit
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Vandetanib | Erlotinib
Number analyzed (Participants) | 623 | 617
Weeks | 11.1 [4.4 to 26] | 9.9 [4.3 to 24.3]

6. Secondary Outcome: Time to Deterioration of Disease-related Symptoms (TDS) by EORTC Quality of Life Questionnaire - Dyspnoea
Description: Dyspnea was assessed as the average score of four items: Question 8 of the QLQ-C30 ("Were you short of breath") and Question 3 of the QLQ-C30 ("Were you short of breath when you rested"), Questions 4 ("Were you short of breath when you walked") and 5 ("Were you short of breath when you climbed stairs") of the QLQ-LC13 (or, equivalently, Questions 33, 34 and 35 of the combined QLQ-C30 and QLQ-LC13 questionnaires).
  Time to deterioration in symptoms is defined as the interval from the date of randomization to the first assessment of worsened without an improvement in the next 28 days. A patient is defined as having a deterioration in symptoms if they have a single visit assessment of 'worsened' with no visit assessment of 'improved' within the next 28 days.
Time Frame: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Vandetanib | Erlotinib
Number analyzed (Participants) | 623 | 617
Weeks | 12 [5.7 to 29.7] | 12.4 [5.1 to 34.4]

7. Secondary Outcome: Time to Deterioration of Disease-related Symptoms (TDS) by EORTC Quality of Life Questionnaire - Cough
Description: Cough was assessed using Question 1 ("How much did you cough") of the QLQ-LC13 (or, equivalently, Question 31 of the combined QLQ-C30 and QLQ-LC13 questionnaires).
  Time to deterioration in symptoms is defined as the interval from the date of randomization to the first assessment of worsened without an improvement in the next 28 days. A patient is defined as having a deterioration in symptoms if they have a single visit assessment of 'worsened' with no visit assessment of 'improved' within the next 28 days.
Time Frame: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Vandetanib | Erlotinib
Number analyzed (Participants) | 623 | 617
Weeks | 15.6 [8.1 to 36.1] | 14.1 [7 to 37.6]

ADVERSE EVENTS:
Description: The Safety Analysis Set included all randomized participant who received at least 1 dose of randomized treatment, 623 in vandetanib and 614 in erlotinib.
Arm/Group | Vandetanib | Erlotinib
Serious Adverse Events (participants affected / at risk) | 197/623 | 155/614
Other Adverse Events (participants affected / at risk) | 539/623 | 542/614
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vandetanib (N=623) | Erlotinib (N=614)
Anaemia (Blood and lymphatic system disorders) | 1 | 5
Febrile Neutropenia (Blood and lymphatic system disorders) | 4 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombotic Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 2 | 0
Atrial Fibrillation (Cardiac disorders) | 2 | 1
Atrial Flutter (Cardiac disorders) | 1 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac Arrest (Cardiac disorders) | 1 | 0
Cardiac Failure (Cardiac disorders) | 2 | 0
Cardio-Respiratory Arrest (Cardiac disorders) | 3 | 0
Cardiopulmonary Failure (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 6 | 2
Pericardial Effusion (Cardiac disorders) | 1 | 0
Postinfarction Angina (Cardiac disorders) | 1 | 0
Right Ventricular Failure (Cardiac disorders) | 1 | 0
Sinus Tachycardia (Cardiac disorders) | 0 | 1
Supraventricular Tachycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Torsade De Pointes (Cardiac disorders) | 1 | 0
Ventricular Fibrillation (Cardiac disorders) | 2 | 0
Ventricular Tachycardia (Cardiac disorders) | 1 | 0
Ulcerative Keratitis (Eye disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 4 | 2
Abdominal Wall Haematoma (Gastrointestinal disorders) | 0 | 1
Colitis Ischaemic (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 19 | 8
Dysphagia (Gastrointestinal disorders) | 4 | 4
Enteritis (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Inguinal Hernia Strangulated (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 5 | 5
Oesophageal Stenosis (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 9 | 9
Asthenia (General disorders) | 4 | 2
Chest Pain (General disorders) | 2 | 1
Chills (General disorders) | 1 | 0
Complication Associated With Device (General disorders) | 0 | 1
Death (General disorders) | 3 | 0
Fatigue (General disorders) | 3 | 4
General Physical Health Deterioration (General disorders) | 3 | 0
Malaise (General disorders) | 0 | 1
Mucosal Inflammation (General disorders) | 1 | 0
Multiple Organ Dysfunction Syndrome (General disorders) | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 0 | 1
Oedema (General disorders) | 0 | 1
Oedema Peripheral (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 7 | 6
Sudden Death (General disorders) | 1 | 3
Biliary Colic (Hepatobiliary disorders) | 1 | 0
Anaphylactic Shock (Immune system disorders) | 1 | 0
Abscess Limb (Infections and infestations) | 1 | 0
Arthritis Bacterial (Infections and infestations) | 1 | 0
Atypical Pneumonia (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 2 | 2
Cellulitis (Infections and infestations) | 1 | 1
Clostridium Colitis (Infections and infestations) | 0 | 1
Conjunctivitis (Infections and infestations) | 1 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Empyema (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis Clostridial (Infections and infestations) | 1 | 0
Genital Infection (Infections and infestations) | 0 | 1
Hepatobiliary Infection (Infections and infestations) | 1 | 0
Herpes Zoster (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 1
Infective Exacerbation Of Chronic Obstructive Airways Disease (Infections and infestations) | 2 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 7 | 6
Lung Infection (Infections and infestations) | 1 | 0
Mycobacterial Infection (Infections and infestations) | 1 | 0
Neutropenic Infection (Infections and infestations) | 1 | 0
Pleural Infection (Infections and infestations) | 0 | 1
Pleural Infection Bacterial (Infections and infestations) | 0 | 1
Pneumococcal Sepsis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 27 | 22
Pneumonia Haemophilus (Infections and infestations) | 0 | 1
Pulmonary Sepsis (Infections and infestations) | 1 | 0
Pulmonary Tuberculosis (Infections and infestations) | 2 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Respiratory Tract Infection (Infections and infestations) | 5 | 4
Sepsis (Infections and infestations) | 1 | 4
Septic Shock (Infections and infestations) | 1 | 1
Streptococcal Bacteraemia (Infections and infestations) | 1 | 0
Subcutaneous Abscess (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 6 | 1
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 2 | 1
Gastroenteritis Radiation (Injury, poisoning and procedural complications) | 0 | 1
Head Injury (Injury, poisoning and procedural complications) | 0 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 1
Radiation Injury (Injury, poisoning and procedural complications) | 0 | 1
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 2 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 | 1
Vascular Graft Occlusion (Injury, poisoning and procedural complications) | 0 | 1
Body Temperature Increased (Investigations) | 0 | 1
C-Reactive Protein Increased (Investigations) | 0 | 2
Electrocardiogram Qt Prolonged (Investigations) | 2 | 0
Electrocardiogram St-T Change (Investigations) | 1 | 0
Electrocardiogram T Wave Inversion (Investigations) | 1 | 0
International Normalised Ratio Increased (Investigations) | 1 | 0
Platelet Count Decreased (Investigations) | 1 | 0
Weight Decreased (Investigations) | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 3 | 4
Dehydration (Metabolism and nutrition disorders) | 7 | 4
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 3
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 3
Spinal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
B-Cell Small Lymphocytic Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4
Lymphangiosis Carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant Pleural Effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Altered State Of Consciousness (Nervous system disorders) | 1 | 1
Aphasia (Nervous system disorders) | 1 | 0
Ataxia (Nervous system disorders) | 0 | 1
Cerebral Infarction (Nervous system disorders) | 0 | 1
Cerebral Ischaemia (Nervous system disorders) | 2 | 0
Cerebral Thrombosis (Nervous system disorders) | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 3
Dizziness (Nervous system disorders) | 3 | 1
Dysarthria (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 0
Hemiparesis (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Paralysis Recurrent Laryngeal Nerve (Nervous system disorders) | 0 | 1
Psychomotor Hyperactivity (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 7 | 3
Somnolence (Nervous system disorders) | 0 | 2
Speech Disorder (Nervous system disorders) | 0 | 1
Spinal Cord Compression (Nervous system disorders) | 0 | 2
Syncope (Nervous system disorders) | 1 | 4
Device Failure (Product Issues) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Completed Suicide (Psychiatric disorders) | 1 | 0
Confusional State (Psychiatric disorders) | 1 | 4
Insomnia (Psychiatric disorders) | 0 | 1
Mental Status Changes (Psychiatric disorders) | 1 | 1
Acute Kidney Injury (Renal and urinary disorders) | 0 | 1
Calculus Urinary (Renal and urinary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 1
Renal Failure (Renal and urinary disorders) | 0 | 1
Tubulointerstitial Nephritis (Renal and urinary disorders) | 1 | 0
Urinary Retention (Renal and urinary disorders) | 1 | 0
Acquired Tracheo-Oesophageal Fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthmatic Crisis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial Fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 | 20
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 11
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pleural Fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 8 | 6
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 0 | 3
Dermatitis Exfoliative (Skin and subcutaneous tissue disorders) | 2 | 0
Eczema Asteatotic (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 7 | 2
Rash Erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash Papular (Skin and subcutaneous tissue disorders) | 0 | 2
Thoracotomy (Surgical and medical procedures) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 1 | 5
Haematoma (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 3 | 1
Hypertensive Crisis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 3
Hypovolaemic Shock (Vascular disorders) | 0 | 1
Jugular Vein Thrombosis (Vascular disorders) | 0 | 1
Orthostatic Hypotension (Vascular disorders) | 0 | 1
Peripheral Arterial Occlusive Disease (Vascular disorders) | 1 | 0
Peripheral Ischaemia (Vascular disorders) | 1 | 0
Subclavian Vein Thrombosis (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vandetanib (N=623) | Erlotinib (N=614)
Constipation (Gastrointestinal disorders) | 58 | 87
Diarrhoea (Gastrointestinal disorders) | 300 | 232
Dyspepsia (Gastrointestinal disorders) | 29 | 31
Nausea (Gastrointestinal disorders) | 138 | 131
Stomatitis (Gastrointestinal disorders) | 33 | 33
Vomiting (Gastrointestinal disorders) | 85 | 91
Asthenia (General disorders) | 50 | 59
Fatigue (General disorders) | 119 | 109
Oedema Peripheral (General disorders) | 21 | 34
Pyrexia (General disorders) | 44 | 50
Paronychia (Infections and infestations) | 12 | 31
Weight Decreased (Investigations) | 33 | 29
Anorexia (Metabolism and nutrition disorders) | 114 | 123
Back Pain (Musculoskeletal and connective tissue disorders) | 37 | 40
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 33 | 24
Dizziness (Nervous system disorders) | 37 | 40
Headache (Nervous system disorders) | 55 | 40
Insomnia (Psychiatric disorders) | 59 | 40
Proteinuria (Renal and urinary disorders) | 33 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 78 | 92
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 84 | 70
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 31 | 39
Acne (Skin and subcutaneous tissue disorders) | 45 | 50
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 75 | 103
Dry Skin (Skin and subcutaneous tissue disorders) | 60 | 84
Pruritus (Skin and subcutaneous tissue disorders) | 38 | 67
Rash (Skin and subcutaneous tissue disorders) | 169 | 232
Hypertension (Vascular disorders) | 99 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.